CLINICAL TRIAL: NCT00278473
Title: Treatment of Meta-Cognitive Deficits in Adults With ADHD
Brief Title: Psychosocial Treatment for Attention Deficit Hyperactivity Disorder in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 03-1059; R34MH071721 (NIH); DATR A2-AIR
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Primarily Inattentive; Hyperactive Impulsive Type; Combined Type; ADHD; Adults; Psychological; Cognitive Behavioral Therapy; CBT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meta-Cognitive Therapy (Experimental): Cognitive behavioral group. Cognitive behavioral therapy focuses on changing patterns of thinking and behavior. Each group consists of 6 to 8 members and sessions are led by a psychologist.
  Interventions: Behavioral: Meta-Cognitive Therapy
- Supportive Therapy (Active Comparator): Social support problem-solving group. Social support problem-solving focuses on general support, problem solving, and information sharing. Each group consists of 6 to 8 members and sessions are led by a psychologist.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Meta-Cognitive Therapy — Cognitive Behavioral Group Treatment
  Other Names: Cognitive Behavioral Group
  Arms: Meta-Cognitive Therapy
Behavioral: Supportive Therapy — Social Support Problem-Solving Group Treatment
  Other Names: Social Support Problem-Solving Group
  Arms: Supportive Therapy

SUMMARY:
This study will determine the effectiveness of group cognitive-behavioral therapy as compared to a problem-solving social support group in treating problems of time management, organization, and planning in adults with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
ADHD is a chronic neurobiological condition that affects people of all ages, genders, and races. Symptoms of ADHD may include, but are not limited to, the following: poor attention span; physical restlessness or hyperactivity; excessive impulsivity; chronic procrastination; frequently losing things; poor organization, planning, and time management skills; and excessive forgetfulness. Not every person with ADHD exhibits all of these symptoms, and the severity of the disorder can range from mild to severe. While there is no cure for ADHD, the condition can be managed with an accurate diagnosis and proper treatment. Left untreated, individuals with ADHD may experience significant impairment in social, emotional, occupational, and academic functioning. Stimulant and non-stimulant medications are usually effective in alleviating symptoms of ADHD in adults. However, some research suggests that medications may not effectively treat self-management functioning problems and that as many as one-third of adults with ADHD have inadequate responses to medication treatment. Additional research on the benefits of psychosocial treatments for ADHD in adults is needed. This study will determine the effectiveness of group cognitive-behavioral therapy as compared to a problem-solving social support group in treating problems of time management, organization, and planning in adults with ADHD.

Individuals interested in participating in this study will first undergo an assessment of their eligibility for inclusion in the study. The assessment will last approximately 6 hours, but can be broken up into as many as 4 separate visits. Eligible participants will be randomly assigned to either receive group cognitive-behavioral therapy or join a problem-solving social support group. Both groups will meet once a week for 12 weeks. Each session will last roughly 2 hours and will focus on building time management, organizational, and planning skills. Time management, planning, and organizational skill levels will be assessed at the treatment mid-point, immediately following the intervention, and at 3 and 6 months following the treatment. Self-esteem and symptoms of depression and anxiety will also be measured at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having or have been diagnosed with ADHD
* May potentially benefit from the ADHD group treatment

Exclusion Criteria:

* Any overt cognitive disability (e.g., Alzheimer's disease, mental retardation)
* Deemed not to potentially benefit from the proposed ADHD group treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary V. Solanto, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participants were referred from New York area medical and psychiatric clinics, ADHD advocacy and self-help groups, community psychiatrists and primary care physicians, university health services, and postings on clinical trials web sites.
Period: Overall Study
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Started | 45 | 43
Completed | 41 | 40
Not Completed | 4 | 3
Not completed — drop out | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.04 (11.59) | 42.37 (12.09) | 41.69 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Inattention Subscale
Description: Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Inattention subscale. Mean change score at 12 weeks as compared to baseline. Each item is scored as follows: 0 (none), 1 (mild), 2 (moderate), 3 (severe); the maximum total score with 27 points being the most severe.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
units on a scale | -13.71 (4.27) | -16.18 (4.71)

2. Primary Outcome: Time Management, Organization, and Planning Subscale
Description: Time management, organization, and planning subscale at posttreatment at 12 weeks as compared to baseline.
  The mean difference On Time Management Organization and Planning scale which is a 24-item self-report questionnaire that uses a 7-point Likert-type scale ranging from -3 (far below average) to +3 (far above average) and subsequently totaled to obtain a composite index of proficiency (possible scores range from -102 to +102), which was developed and previously used at the ADHD program at the Icahn School of Medicine at Mount Sinai.
Time Frame: baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
units on a scale | -7.66 (2.83) | -9.70 (3.16)

3. Secondary Outcome: CAARS-O:L
Description: Change in the Conners Adult ADHD Rating Scales-Observer: Long Version (CAARS-O:L), inattention/memory subscale at 12 weeks as compared to baseline. 12 items subscale. T-score of at least 63 gives risk or possible diagnosis of ADHD. This number, lower or higher, does not indicate severity.
Time Frame: baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
T-score | -66.94 (11.64) | -73.19 (10.33)

4. Secondary Outcome: Beck Depression Inventory
Description: Mean change in the Beck Depression Inventory Scale at 12 weeks as compared to baseline.
  The Beck Depression Inventory, 2nd edition to assess Depression symptoms. BDI-II scores range between 0 and 63, with categorical depression ratings of "minimal" (0-13), "mild" (14-19), "moderate" (20-28), and "severe" (29-63).
Time Frame: baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
units on a scale | -9.66 (8.31) | -9.08 (7.16)

5. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: Mean Change in Hamilton Anxiety Rating Scale at 12 weeks as compared to baseline. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
units on a scale | -8.07 (5.38) | -8.88 (5.63)

6. Secondary Outcome: Rosenberg Self-Esteem Inventory
Description: Mean change in Rosenberg Self-Esteem Inventory score at 12 weeks as compared to baseline. The scale is a ten item Likert scale, ranging from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
Time Frame: baseline and at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Number analyzed (Participants) | 41 | 40
units on a scale | -18.39 (6.02) | -19.5 (5.86)

ADVERSE EVENTS:
Description: Adverse effects information not collected
Arm/Group | Meta-Cognitive Therapy | Supportive Therapy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
participants were required to meet minimum levels of severity of symptoms and may select nonresponders or suboptimal responders to medication.

Small sample may affects potential moderating and mediating variables

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes